CLINICAL TRIAL: NCT03848143
Title: Intraoral Administration of Onabotulinum Toxin A for Continuous Neuropathic Pain: a Single Subject Experimental Design
Brief Title: Intraoral Administration of Botox in Patients With Dentoalveolar Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isabel Moreno Hay (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Isabel Moreno Hay, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 45231; IIT-10247 (Other: Allergan Sales LLC)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Single subject experimental design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BOTOX (Experimental): Onabotulinum toxin A is distributed in 50 unit (50U) vacuum-dried powder bottles by Allergan (BOTOX (R)) for reconstitution only with sterile, preservative-free 0.9% Sodium Chloride Injection prior to injection.
  1 mL of diluent will be drawn up to obtain a resulting dose of 10 U per 0.2 mL and injected into the vial. The BOTOX(R) will then be gently mixed with the saline by rotating the vial. The date and time of reconstitution will be recorded on the package on the label. BOTOX should be administered within 24 hours after reconstitution and stored in a refrigerator (2-8 °C).
  Each patient will receive 50 U of onabotulinum toxin A.
  Interventions: Drug: onabotulinum toxin A

INTERVENTIONS:
Drug: onabotulinum toxin A — Each subject will receive 50 units (50 U) of BoNT-A constituted in 1 mL of saline solution injected intraorally to the painful area divided in at least 3 sites, 0.5 to 1.0 cm apart depending on the size of the painful area and following a checkerboard pattern.
  Other Names: BOTOX

SUMMARY:
Onabotulinum toxin type A (BoNT-A) is a potent neurotoxin that has been reported to have an effect on afferent (sensory) neurons independent of its action on muscle tone and secretory glands at the periphery.In human studies, the use of BoNT-A has proven to reduce the severity and intensity of attacks in chronic tension type headaches and chronic neck pain. The PREEMPT study concluded that BoNT-A could be used as a preventive therapy in chronic migraine patients and FDA approval was obtained. According to the International Association for the Study of Pain (IASP), BoNT-A is recommended for the management of peripheral neuropathic pain with subcutaneous administration of 50-200 units (50-200U) to onabotulinum toxin A to the painful neuropathic area every 3 months as a third line of treatment. To our knowledge, there are no clinical trials published investigating the effect of intraoral administration of BoNT-A in continuous dentoalveolar neuropathic pain. The aim of this pilot study is to investigate the potential therapeutic effect of intraoral administration of BoNT-A in patients suffering from continuous neuropathic pain.

HYPOTHESIS:

There will be statistically significant differences in reported pain intensity after the intraoral administration of BOTOX® in patients suffering from chronic continuous dentoalveolar neuropathic pain.

A single subject experiment will be conducted with 10 patients where 50 U of BonT-A will be injected into the painful dentoalveolar area. Eligible subjects will complete a pain diary indicating their pain intensity by means of a visual analog scale during one month to establish a baseline. After the first injection, subjects will continue to monitor the VAS daily for 3 months and the infiltration will be repeated a second time following the same protocol. Patient's response will be monitored with the daily pain diary.

ELIGIBILITY:
Inclusion Criteria:

* History of continuous dentoalveolar pain with clinically evident positive (hyperalgesia, allodynia) and/or negative (hypoaesthesia, hypoalgesia) signs of trigeminal nerve dysfunction and where other possible pain sources have been ruled out.
* Intractable pain to conventional oral and/or topical pharmacotherapy for neuropathic pain according to the recommendations published by NeuPSIG (Neuropathic Pain Special Interest Group) including anticonvulsants, SNRIs (serotonin and norepinephrine reuptake inhibitors) and/or tricyclic antidepressants.
* Subject consent to participate in the study.

Exclusion Criteria:

* hypersensitive to any onabotulinum toxin preparation or any component in the formulation.
* systemic nerve or muscle disorders
* bleeding disorders
* dysphagia
* breathing problems
* pregnancy or breastfeeding
* previous treatment with botulinum toxin in the last 4 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Over 7 months
  Patient will record the pain intensity by means of a visual analogue scale (VAS, from 0-10 being 0 no pain and 10 the worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Okeson, DMD, Study Director — Associate Professor
Locations (1):
- Orofacial Pain Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolly JO, O'Connell MA. Neurotherapeutics to inhibit exocytosis from sensory neurons for the control of chronic pain. Curr Opin Pharmacol. 2012 Feb;12(1):100-8. doi: 10.1016/j.coph.2011.11.001. Epub 2011 Dec 19. PMID 22188874
- [Background] Cui M, Khanijou S, Rubino J, Aoki KR. Subcutaneous administration of botulinum toxin A reduces formalin-induced pain. Pain. 2004 Jan;107(1-2):125-33. doi: 10.1016/j.pain.2003.10.008. PMID 14715398
- [Background] Luvisetto S, Marinelli S, Lucchetti F, Marchi F, Cobianchi S, Rossetto O, Montecucco C, Pavone F. Botulinum neurotoxins and formalin-induced pain: central vs. peripheral effects in mice. Brain Res. 2006 Apr 12;1082(1):124-31. doi: 10.1016/j.brainres.2006.01.117. Epub 2006 Mar 9. PMID 16524562
- [Background] Bach-Rojecky L, Lackovic Z. Antinociceptive effect of botulinum toxin type a in rat model of carrageenan and capsaicin induced pain. Croat Med J. 2005 Apr;46(2):201-8. PMID 15849840
- [Background] Marinelli S, Luvisetto S, Cobianchi S, Makuch W, Obara I, Mezzaroma E, Caruso M, Straface E, Przewlocka B, Pavone F. Botulinum neurotoxin type A counteracts neuropathic pain and facilitates functional recovery after peripheral nerve injury in animal models. Neuroscience. 2010 Nov 24;171(1):316-28. doi: 10.1016/j.neuroscience.2010.08.067. Epub 2010 Sep 6. PMID 20826198
- [Background] Bach-Rojecky L, Relja M, Lackovic Z. Botulinum toxin type A in experimental neuropathic pain. J Neural Transm (Vienna). 2005 Feb;112(2):215-9. doi: 10.1007/s00702-004-0265-1. PMID 15657640
- [Background] Park HJ, Lee Y, Lee J, Park C, Moon DE. The effects of botulinum toxin A on mechanical and cold allodynia in a rat model of neuropathic pain. Can J Anaesth. 2006 May;53(5):470-7. doi: 10.1007/BF03022619. PMID 16636031
- [Background] Bach-Rojecky L, Salkovic-Petrisic M, Lackovic Z. Botulinum toxin type A reduces pain supersensitivity in experimental diabetic neuropathy: bilateral effect after unilateral injection. Eur J Pharmacol. 2010 May 10;633(1-3):10-4. doi: 10.1016/j.ejphar.2010.01.020. Epub 2010 Feb 1. PMID 20123097
- [Background] Filipovic B, Bach-Rojecky L, Lackovic Z. Lasting reduction of postsurgical hyperalgesia after single injection of botulinum toxin type A in rat. Fundam Clin Pharmacol. 2010 Feb;24(1):43-5. doi: 10.1111/j.1472-8206.2009.00767.x. Epub 2009 Aug 14. PMID 19682079
- [Background] Relja M, Telarovic S. Botulinum toxin in tension-type headache. J Neurol. 2004 Feb;251 Suppl 1:I12-4. doi: 10.1007/s00415-004-1104-x. PMID 14991337
- [Background] Miller D, Richardson D, Eisa M, Bajwa RJ, Jabbari B. Botulinum neurotoxin-A for treatment of refractory neck pain: a randomized, double-blind study. Pain Med. 2009 Sep;10(6):1012-7. doi: 10.1111/j.1526-4637.2009.00658.x. Epub 2009 Jul 6. PMID 19594841
- [Background] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710